CLINICAL TRIAL: NCT06260709
Title: Open-label Extension Study of Long-term Safety and Efficacy of NNC6019-0001 in Participants With Transthyretin Amyloid Cardiomyopathy (ATTR CM)
Brief Title: A Research Study to Look at Long-term Treatment With a Medicine Called NNC6019-0001 for People Who Have Heart Failure Due to Transthyretin Amyloidosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN6019-7565; 2022-502605-15-00 (Other: European Medical Agency (EMA)); U1111-1284-5820 (Other: World Health Organization (WHO)); jRCT2071240078 (Registry Identifier: JRCT)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Transthyretin Amyloid Cardiomyopathy (ATTR CM)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNC6019-0001 (Experimental): Participants will receive NNC6019-0001 intravenously every 4 weeks added to the standard of care until Week 140.
  Interventions: Drug: NNC6019-0001

INTERVENTIONS:
Drug: NNC6019-0001 — Intravenous NNC6019-0001 every 4 weeks added to the standard of care until Week 140.

SUMMARY:
This study will test a medicine, NNC6019-0001, for people who have a heart disease due to TTR amyloidosis. It will look at how safe this medicine is in the long term and if it can reduce symptoms of a heart disease due to TTR amyloidosis, such as heart failure. It is an extension to a study called "A research study to look at how a new medicine called NNC6019-0001 works and how safe it is for people who have a heart disease due to TTR amyloidosis". Only participants who have completed that study will be invited for this new study. Participants will get NNC6019-0001, regardless of whether they got placebo or NNC6019-0001 in the first study. The study will last for up to 157 weeks (36 months/3 years).

ELIGIBILITY:
Inclusion Criteria:

* Completed study intervention in NN6019-4940 and attended the last study visit (week 64; visit 16), and no later than 12 weeks after visit 16.
* Expected to be on stable doses of cardiovascular medical therapy 6 weeks prior to the enrolment visit.

Exclusion Criteria:

* A prior solid organ transplant.
* Presence or history of malignant neoplasm (other than basal or squamous cell skin cancer, in-situ carcinomas of the cervix, or in-situ/high grade prostatic intraepithelial neoplasia (PIN) or low-grade prostate cancer) within 5 years before screening.
* Current treatment with calcium channel blockers with conduction system effects (e.g., verapamil, diltiazem). The use of dihydropyridine calcium channel blockers is allowed. The use of digoxin will only be allowed if required for management of atrial fibrillation with rapid ventricular response.
* Body weight greater than (>) 120 kilograms (kg) (264.6 pounds [lb]) at screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment Emergent Adverse Events | From baseline (week 0) up to visit 39 (week 156)
  Measured as events.

SECONDARY OUTCOMES:
Change in 6-Minute Walk Test (6MWT) | From baseline (week 0) to visit 28 (week 104)
  Measured in meters.
Change in N-terminal-pro brain natriuretic peptide (NT-proBNP) | From baseline (week 0) to visit 28 (week 104)
  Measured in percentage.
Change in Myocardial Extracellular Volume (ECV) | From baseline (week 0) to visit 28 (week 104)
  Measured in percentage-points.
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score (CSS) | From baseline (week 0) to visit 28 (week 104)
  The KCCQ is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and health-related quality of life limitation from heart failure. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. CSS scores range from 0 to 100 and lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life. Measured in score on a scale.
Change in Troponin I | From baseline (week 0) to visit 28 (week 104)
  Measured in nanogram per milliliter (ng/mL).
Change in Global Longitudinal Strain (GLS) on Echocardiography | From baseline (week 0) to visit 28 (week 104)
  Measured in percentage-points.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (35):
- United States (8):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Cedars-Sinai Medical Center_Los Angeles, Los Angeles, California
  - Stanford Hlth Cre-Boswell Clin, Stanford, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - NW Univ-Bluhm Cardiovasc Inst, Chicago, Illinois
  - NW Univ-Bluhm Cardiovasc Inst, Evanston, Illinois
  - Univ of MD Schl of Med, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
- Canada (2):
  - University of Calgary_Cardiology, Calgary, Alberta
  - Ctr for Cardiovascular Innovation, Vancouver, British Columbia
- II. interni klinika VFN - Kardiologie a angiologie, Prague, Czechia
- France (2):
  - Ap-Hp-Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-1, Toulouse
- Germany (7):
  - UniklinikHeidelberg - Innere Med. III - Kardiologie, Angiologie, Pneumologie, Heidelberg
  - Universitätsklinik Heidelberg Innere Medizin III Kardiologie, Angiologie, Pneumologie, Heidelberg
  - LMU Klinikum München Klinik und Poliklinik 1, München
  - Uniklinik Münster, Klinik für Kardiologie I, Münster
  - Universitätsklinikum Münster - Klinik für Kardiologie I, Münster
  - Universitatsklinikum Wurzburg AöR, Würzburg
  - Universitatsklinikum Würzburg - Zentrum für Herzinsuffizienz, Würzburg
- Italy (3):
  - Fondazione CNR-Regione Toscana Gabriele Monasterio, Pisa, Pi
  - Fondazione Toscana Gabriele Monasterio - Dipartimento Cardiotoracico - UOC Cardiologia e Medicina Cardiovascolare, Pisa, Pi
  - Centro per lo Studio e la Cura delle Amiloidosi Sistemiche Fondazione IRCCS Policlinico San Matteo, Pavia, PV
- Japan (6):
  - Hospital of the University of Occupational and Environmental Health, Cardiology, Nephrology, Fukuoka
  - Hiroshima University hospital, Cardiovascular Medicine, Hiroshima
  - Kumamoto University Hospital, Cardiovascular Medicine, Kumamoto-shi, Kumamoto
  - Shinshu University Hospital, Department of Neurology, Nagano
  - Nagasaki University Hospital, Cardiovascular Medicine, Nagasaki
  - Okayama University Hospital_Cardiovascular Medicine, Okayama-shi, Okayama
- Netherlands (2):
  - UMC Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Portugal (3):
  - Hospital da Senhora da Oliveira - Guimarães, Guimarães
  - Unidade Local de Saude do Alto Ave, E.P.E., Guimarães
  - Unidade Local De Saude De Tras-Os-Montes E Alto Douro E.P.E., Vila Real
- Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com